CLINICAL TRIAL: NCT01434186
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Saxagliptin (BMS-477118) in Combination With Metformin IR or Metformin XR in Pediatric Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-147; 2010-024568-16 (EudraCT Number)
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Saxagliptin +Metformin XR/IR (Experimental): Saxagliptin Tablet, 2.5 mg, or Saxagliptin Tablet, 5 mg, (based on subject's weight) Metformin XR/IR 1000 mg-2000 mg
  Interventions: Drug: Metformin IR; Drug: Metformin XR; Drug: Saxagliptin
- Arm 2: Placebo +Metformin XR/IR (Placebo Comparator): Placebo matching saxagliptin 0 mg Metformin XR/IR 1000 mg - 2000 mg
  Interventions: Drug: Placebo matching with Saxagliptin; Drug: Metformin IR; Drug: Metformin XR

INTERVENTIONS:
Drug: Placebo matching with Saxagliptin — Tablet, Oral, 0.0 mg, Daily, Day 1 through week 52
  Arms: Arm 2: Placebo +Metformin XR/IR
Drug: Metformin IR — Tablet, Oral, 1000 mg -2000 mg, Daily , Day 1 through week 52
Drug: Metformin XR — Tablet, Oral, 1000 mg -2000 mg, Daily, Day 1 through week 52
Drug: Saxagliptin — Saxagliptin Tablet, 2.5 mg, or Saxagliptin Tablet, 5 mg, (based on subject's weight)
  Other Names: BMS-477118
  Arms: Arm 1: Saxagliptin +Metformin XR/IR

SUMMARY:
To evaluate the efficacy, safety, tolerability, of Saxagliptin (BMS-477118) in combination with Metformin in pediatric patients with type 2 diabetes

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Saxagliptin (BMS-477118) in Combination with Metformin IR or Metformin XR in Pediatric Patients with Type 2 Diabetes who have Inadequate Glycemic Control on Metformin Alone or in Combination with Baseline Insulin Therapy

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients eligible if 10 years of age, up to 17 years and 30 weeks of age at the time of screening
* Previously diagnosed as having type 2 diabetes
* HbA1c ≥7.0% and ≤10.5%
* Body weight ≥ 30 kg
* Stable dose of metformin (≥ 1000mg - ≤ 2000mg) for a minimum of 2 months
* Women must have a negative serum or urine pregnancy test
* Women must not be breastfeeding

Exclusion Criteria:

* Current use of anti-diabetic medications or use within the specified timeframe prior to screening (Exception: Metformin)
* Fasting plasma glucose (FPG) > 255 mg/dL
* Diabetic ketoacidosis (DKA) within 6 months of study entry
* Abnormal renal function
* Active liver disease
* Anemia
* An abnormal Thyroid Stimulating Hormone (TSH)
* Creatinine kinase (CK) ≥ 3X ULN

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Tallahassee, Florida
  - Research Site, Dearborn, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, Mineola, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Memphis, Tennessee
- Research Site, Namur, Belgium
- Research Site, Calgary, Alberta, Canada
- Research Site, Bangalore, India
- Mexico (4):
  - Research Site, Aguascalientes
  - Research Site, Meridas
  - Research Site, Monterrey
  - Research Site, Veracruz
- Research Site, Taichung, Taiwan
- Research Site, Leicester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 32 subjects enrolled, 7 subjects entered the lead-in period. Of these 7 subjects, 6 were randomized
Groups:
- Placebo: Placebo matching saxagliptin
- Saxagliptin: saxagliptin 2.5 or 5 mg according to body weight
Period: Overall Study
Arm/Group | Placebo | Saxagliptin
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Saxagliptin | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 4 | 6
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in HbA1c From Baseline to Week 16
Time Frame: 16 week short term treatment period
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Saxagliptin: Saxagliptin 2.5 mg or 5 mg according to bodyweight
- Placebo: Saxagliptin matching placebo
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 4 | 2
percentage | -1.0 (0.62) | 0.9 (0.14)

ADVERSE EVENTS:
Time Frame: 52 week
Arm/Group | Placebo | Saxagliptin
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 1/2 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | Saxagliptin (N=4)
Headache (Nervous system disorders) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngitis Streptococcal (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis bacterial (Infections and infestations) | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 1 | 0
URINE OUTPUT INCREASED (Investigations) | 1 | 0
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No